CLINICAL TRIAL: NCT02594241
Title: PreOperative Steroid in Abdominal Wall Reconstruction: A Double-blinded Randomized Clinical Trial
Acronym: POSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Kiim Jensen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kiim Jensen, MD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-806
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Hernia, Ventral
Keywords: Ventral hernia; Abdominal wall reconstruction; Enhanced recovery after surgery; Steroid
MeSH Terms: conditions — Hernia, Ventral | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Patients in this arm will be given an intravenous infusion of 125 mg Methylprednisolone (Solu-Medrol) immediately after induction of general anesthesia.
  Interventions: Drug: Methyl-Prednisolone
- Physiological saline (Placebo Comparator): Patients in this arm will be given an intravenous infusion of saline immediately after induction of general anesthesia.
  Interventions: Drug: Physiological saline

INTERVENTIONS:
Drug: Methyl-Prednisolone — Single-shot 125 mg infusion given immediately after induction of anesthesia.
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Physiological saline — A single preoperative dosage 100 ml given intravenously as a 30 minute infusion, 2 hours before surgery
  Other Names: Physiological Saline 9 mg/ml, Fresenius Kabi
  Arms: Physiological saline

SUMMARY:
Patients who undergo abdominal wall reconstruction for giant ventral hernia repair will be randomized to either methylprednisolone or saline preoperatively, to examine the effects of methylprednisolone on postoperative pain, nausea and recovery after giant ventral hernia repair.

DETAILED DESCRIPTION:
Preoperative high-dose glucocorticoid has been shown to attenuate the postoperative inflammatory response leading to decreased morbidity and length of stay (LOS) after colorectal and aortic surgery, as well as decreased pain and subjective recovery after orthopedic surgery. Methylprednisolone (MP, "Solu-Medrol") is one such glucocorticoid, which has been shown to be safe for usage in surgery. Giant ventral hernia repair is associated with a high risk of postoperative morbidity and prolonged LOS compared with other hernia repair procedures requiring laparotomy. Further, the total costs of these procedures remain high. Systemic administration of high-dose preoperative MP in ventral hernia repair has only been described anecdotally in the literature, and never with the aim to improve the treatment of this patient group specifically. It is however unknown to what extent benefits weigh out downsides from usage of high-dose MP in giant ventral hernia repair, patients often at increased risk of postoperative wound infection. On this background we hypothesize that a preoperative high-dose MP results in improved recovery after giant ventral hernia repair compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ventral incisional hernia with horizontal fascial defect > 10 cm described at either computed tomography scan or clinical assessment
* Planned elective open hernia repair
* Ability to speak and understand Danish
* Ability to give written and oral informed consent

Exclusion Criteria:

* Daily use of systemic glucocorticoid
* New York Heart Association class 3-4 heart disease
* Chronic renal failure (eGFR < 60 ml/min per 1.73 m2)
* Insulin-dependent diabetes
* Excessive abuse of alcohol
* Known allergy to methylprednisolone or any substance in study medicine
* Planned pregnancy within three months postoperatively
* Pregnancy, evaluated by pregnancy test preoperatively
* Breastfeeding
* Actively treated ulcer disease up to one month preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Pain at rest | First postoperative day at 8 am
  Self-reported pain at rest on af numerical rating scale (0-10)

SECONDARY OUTCOMES:
Pain at rest, after moving from supine to sitting position and when coughing | 8 am and 8 pm pre- and postoperatively until postoperative day 5 and again on day 30
  Self-reported pain at rest, after moving from supine to sitting position and when coughing on af numerical rating scale (0-10)
Fatigue | 8 am and 8 pm pre- and postoperatively until postoperative day 5 and again on day 30
  Self-reported fatigue on a numerical rating scale (0-10)
Nausea | 8 am and 8 pm pre- and postoperatively until postoperative day 5 and again on day 30
  Self-reported nausea on a numerical rating scale (0-10)
Vomiting | From randomization until postoperative day 5
  Number of vomiting episodes
Time to fulfillment of discharge criteria | From randomization until postoperative day 5, assessed at 8 am and 8 pm
  Patient's assessment of discharge criteria
30-postoperative complications | From randomization and until 30-days postoperatively
  Complications that require surgical or medical intervention
30-day readmission | From randomization and until 30-days postoperatively
  Patient readmission
Rescue analgesia intake | From randomization and until day 5 postoperatively
  Need for intake of rescue analgesia postoperatively
C-reactive protein | From day of randomization until postoperative day 3
  Serum C-reactive protein preoperatively and on postoperative day 1-3.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Jensen, MD, Principal Investigator — Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark

REFERENCES:
- [Derived] Jensen KK, Brondum TL, Belhage B, Hensler M, Arnesen RB, Kehlet H, Jorgensen LN. Preoperative steroid in abdominal wall reconstruction: protocol for a randomised trial. Dan Med J. 2016 Aug;63(8):A5260. PMID 27477797